CLINICAL TRIAL: NCT01941745
Title: Efficacy of Recombinant Human Clara Cell Protein (rhCC10) Administered to Premature Neonates With Respiratory Distress Syndrome
Brief Title: Efficacy of Recombinant Human Clara Cell 10 Protein (rhCC10) Administered to Premature Neonates With Respiratory Distress Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tufts Medical Center (Other)
Collaborators: Brigham and Women's Hospital (Other); Therabron Therapeutics, Inc. (Industry); Baystate Medical Center (Other); Poznan University of Medical Sciences (Other); SP ZOZ Szpital Uniwersytecki w Krakowie Oddizat Neonatologii (Unknown); Instytut Centrum Zdrowia Matki Polki Klinika Neonatologii (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: rhCC10 Study 2013; Grant #3899 (Other Grant/Funding Number: FDA OOPD)
Record Dates: First submitted 2013-08-29; First posted 2013-09-13 (Estimated); Results first posted 2019-09-10 (Actual); Last update posted 2019-09-10 (Actual); Status verified 2019-08

CONDITIONS: Respiratory Distress Syndrome in Premature Infant; Bronchopulmonary Dysplasia
MeSH Terms: conditions — Bronchopulmonary Dysplasia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- half normal saline (Placebo Comparator): Single dose of half normal saline at 2 ml/kg given intratracheally times one dose
  Interventions: Drug: Half normal saline
- Low Dose rhCC10 (Experimental): 1.5 mg/kg study drug (rhCC10)in 2 ml/kg given intratracheally times one dose
  Interventions: Drug: Low Dose rhCC10
- High dose rhCC10 (Experimental): 5 mg/kg of rhCC10 given in 2 ml/kg and administered intratracheally times one dose
  Interventions: Drug: High dose rhCC10

INTERVENTIONS:
Drug: Half normal saline — 2 ml/kg
  Arms: half normal saline
Drug: Low Dose rhCC10 — 1.5 mg/kg study drug (rhCC10)
  Arms: Low Dose rhCC10
Drug: High dose rhCC10 — 5 mg/kg in 2 ml/kg
  Arms: High dose rhCC10

SUMMARY:
Bronchopulmonary Dysplasia (BPD) is a multi-factorial disease process that is the end result of an immature, surfactant deficient lung that has been exposed to hyperoxia, mechanical ventilation and infection. These conditions initiate an inflammatory response characterized by elevated inflammatory cell infiltrates and proinflammatory cytokines that lead to the development of significant acute and chronic lung injury.

The study drug, rhCC10, is a recombinant version of natural human CC10 protein. Native CC10 is produced primarily by non-ciliated respiratory epithelial cells, called Clara cells and is the most abundant protein in the mucosal fluids in normal healthy lungs.

The purpose of this study is to evaluate the pharmacokinetics, safety, tolerability and anti-inflammatory effects of a single intratracheal (IT) dose of rhCC10 to intubated premature infants receiving positive pressure ventilation for treatment of respiratory distress syndrome (RDS) to prevent long term respiratory complications referred to as bronchopulmonary dysplasia, and, more recently, as Chronic Pulmonary Insufficiency of Prematurity (CPIP; asthma, cough, wheezing, multiple respiratory infections).

CC10 regulates inflammatory responses and protects the structural integrity of pulmonary tissue while preserving pulmonary mechanical function during various insults (eg. viral infection, bacterial endotoxin, ozone, allergens, hyperoxia). Together these properties suggest that administration of rhCC10 may help to facilitate development of normal airway epithelia and prevent the inflammation that leads to CPIP in these infants.

This study is funded by the FDA Office of Orphan Product Development (OOPD).

DETAILED DESCRIPTION:
Recombinant human CC10 protein (rhCC10) is a novel therapeutic agent used to prevent the development of chronic respiratory morbidity (CPIP; repeated respiratory infections, asthma, re-hospitalizations) in preterm infants. Native CC10 is a natural anti-inflammatory and immunomodulatory factor produced by Clara Cells in the lung and is the most abundant protein in respiratory mucosa. Animal data demonstrate that a single intratracheal dose of rhCC10 administered shortly after birth reduces lung inflammation (important biomarkers linked to lung injury in preterm infants), promotes normal lung development, preserves lung architecture, improves pulmonary function, suppresses the response to endotoxin and enhances resistance to pulmonary infections. In preterm infants who die or develop lung inflammation and subsequent bronchopulmonary dysplasia (BPD), both the concentration and activity of CC10 are significantly reduced indicating that CC10 is essential for preventing lung injury and promoting normal lung development. In a small phase I study, rhCC10 significantly decreased several indices of pulmonary inflammation in the lungs of premature infants who were at risk of developing BPD and associated CPIP. The drug appeared to be safe, well-tolerated, and reduce risk of re-hospitalization due to respiratory illness for 9-10 months after a single intratracheal dose at the time of birth (0/11 rhCC10-treated infants vs. 3/6 placebo-treated). This supports the protective role of rhCC10 against damage from hyperoxia, mechanical ventilation, inflammation, and infection in the immature lung. A more normal airway epithelium will produce significantly more endogenous CC10, with both factors contributing to enhanced resistance to infections, less asthma, and improved long-term respiratory outcome. We propose to conduct a Phase 2 clinical trial to evaluate rhCC10 in extremely premature infants (<29 weeks gestation) for the prevention of BPD and CPIP. This will be a randomized, double-blind, placebo-controlled dose escalation study in 88 premature infants. A single intratracheal dose of study drug (rhCC10 or placebo) will be administered to preterm infants receiving surfactant and mechanical ventilation for treatment of RDS. Infants will be followed to evaluate safety, pharmacokinetics, and short and long term efficacy of this approach. Safety will be evaluated through serious adverse event (SAE) and adverse event monitoring and by Bayley neurodevelopmental assessments at 18 months corrected gestational age (CGA). Efficacy measurements will include the primary combined endpoint of alive without evidence of CPIP through 12 months CGA (defined by parental diaries and pulmonary questionnaires) comparing rhCC10 treated to placebo controls. The availability of a therapy which prevents lung injury, promotes lung development, and prevents serious respiratory infections and asthma in high risk preterm infants would be a highly significant advancement in care.

ELIGIBILITY:
Inclusion Criteria:

* Age less than or equal to 24 hours;
* Birth weight 600 - 1250 grams;
* Gestational age 24-29 weeks (not less than 24 weeks); at birth based on best estimate using obstetrical sonography (first or second trimester), solid dating criteria, or Ballard examination;
* Birth weight appropriate for gestational age;
* 5 minute Apgar score >5;
* Diagnosis of neonatal RDS based on clinical and radiographic criteria;
* Requiring intubation and mechanical ventilation for treatment of RDS;
* Received at least one dose of surfactant (prophylaxis or rescue); and
* Written informed consent is obtained from at least one of the infant's parents or legal guardians (see section 6.2) prior to enrollment of the subject. The parent(s) or legal guardian(s) must agree to all study-related procedures and evaluations.

Exclusion Criteria:

* 5 minute Apgar score of ≤ 5;
* Major congenital anomaly (chromosomal, renal, cardiac, hepatic, neurologic, or pulmonary malformations; minor anomalies such as cleft lip/palate are permitted);
* Evidence of severe neonatal depression (as defined by cord blood acid-base balance (pH) ≤ 7.00 and/or an Apgar score of < 4 at 10 minutes);
* Evidence of congenital infection;
* Requires a major surgical procedure prior to administration of Study drug
* Enrollment in any other study involving administration of another investigational drug;
* Any condition which could preclude receiving study drug or performing any study-related procedures;
* Use of postnatal corticosteroids prior to administration of r-hCC10, except as specified in the protocol;
* Use of inhaled nitric oxide prior to administration of r-hCC10;
* Mother is known to be seropositive for HIV (per maternal medical records);
* Parent or guardian is unable or unwilling to complete the study diary;
* Parent or guardian is unable to bring the infant back to the study center for follow-up evaluations.

Ages: 24 Weeks to 29 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 88 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2017-08-25 (Actual); Study Completion 2017-08-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Davis, MD, Principal Investigator — Tufts Medical Center; Richard Parad, MD/MPH, Principal Investigator — Brigham and Women's Hospital
Locations (3):
- United States (3):
  - Tufts Medical Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment spanned October 2013 - August 2017 at ICUs at Tufts Medical Center (Boston, MA), Brigham and Women's Hospital (Boston, MA), and BayState Medical Center (Springfield, MA). Three hospital sites in Poland were later added for the second high-dose/high dose placebo cohort of 44 neonates.
Pre-assignment Details: No washout/run-in events to report.
Groups:
- Placebo (Associated w/ Low Dose Cohort): Dosage: Single dose of half normal saline at 2 ml/kg
  Administration: once intratracheally within the first 24 hours of life, and once within 4 hours of the first dose of exogenous surfactant (CurosurfTM)
  Enrollment: 22 participants
- Low Dose (rhCC10): Dosage: 1.5 mg/kg study drug rhCC10 in 2 ml/kg
  Administration: once intratracheally within the first 24 hours of life, and once within 4 hours of the first dose of exogenous surfactant (CurosurfTM)
  Enrollment: 22 participants
- Placebo (Associated w/ High Dose Cohort): Dosage: Single dose of half normal saline at 2 ml/kg
  Administration: once intratracheally within the first 24 hours of life, and once within 4 hours of the first dose of exogenous surfactant (CurosurfTM)
  Enrollment: 21 participants
- High Dose (rhCC10): Dosage: 5 mg/kg of rhCC10 given in 2 ml/kg
  Administration: once intratracheally within the first 24 hours of life, and once within 4 hours of the first dose of exogenous surfactant (CurosurfTM)
  Enrollment: 23 participants
Period: Overall Study
Arm/Group | Placebo (Associated w/ Low Dose Cohort) | Low Dose (rhCC10) | Placebo (Associated w/ High Dose Cohort) | High Dose (rhCC10)
Started | 22 | 22 | 21 | 23
Completed | 22 | 22 | 21 | 23
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline populations were recruited from Tufts Medical Center and Brigham and Women's Hospital. Sites with a second high-dose cohort include BayState Medical Center, Ginekologiczno-Położniczy Szpital Kliniczny UM, Instytut Centrum Zdrowia Matki Polski and Samodzielny Publiczny Zakład Opieki Zdrowotnej Szpital Uniwersytecki w Krakowie (US, Poland).
Groups:
- Placebo (Associated w/ High Dose Cohort): Dosage: Single dose of half normal saline at 2 ml/kg
  Administration: once intratracheally within the first 24 hours of life, and once within 4 hours of the first dose of exogenous surfactant (CurosurfTM)
  Enrollment: 23 participants
- Total: Total of all reporting groups
Arm/Group | Placebo (Associated w/ Low Dose Cohort) | Low Dose (rhCC10) | Placebo (Associated w/ High Dose Cohort) | High Dose (rhCC10) | Total
Number analyzed (Participants) | 22 | 22 | 21 | 23 | 88
Age, Customized [Mean (Standard Deviation); unit: weeks] — Mean gestational age at birth (in weeks, SD)
  weeks | 26.1 (1.3) | 26.5 (1.1) | 27.0 (1.3) | 26.6 (1.2) | 26.6 (1.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 8 | 8 | 12 | 40
  Male | 10 | 14 | 13 | 11 | 48
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Hispanic/Latino or unknown ethnicity by number of participants, n (%).
  Participants
    Hispanic or Latino | 5 | 7 | 5 | 5 | 22
    Not Hispanic or Latino | 0 | 0 | 0 | 0 | 0
    Unknown or Not Reported | 17 | 15 | 16 | 18 | 66
Race (NIH/OMB) [Count of Participants; unit: Participants] — Number of participants, N(%)
  Participants
    American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
    Asian | 0 | 0 | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
    Black or African American | 0 | 0 | 0 | 0 | 0
    White | 9 | 12 | 15 | 18 | 54
    More than one race | 0 | 0 | 0 | 0 | 0
    Unknown or Not Reported | 13 | 10 | 6 | 5 | 34
Region of Enrollment [Number; unit: participants] — Count of participants enrolled in the US (Tufts Medical Center, Brigham and Women's Hospital, Bay State Medical Center) and Poland (Ginekologiczno-Położniczy Szpital Kliniczny UM, Instytut Centrum Zdrowia Matki Polski, and Samodzielny Publiczny Zakład Opieki Zdrowotnej Szpital Uniwersytecki w Krakowie). All three sites in Poland administered the high dose CC10/placebo cohorts only.
  participants
    United States | 22 | 22 | 10 | 11 | 65
    Poland | 0 | 0 | 11 | 12 | 22
Mean birth weight [Mean (Standard Deviation); unit: grams] — in grams (SD)
  grams | 877.4 (170.9) | 859.3 (140.9) | 885.5 (173.9) | 867.2 (187.2) | 874.5 (168.2)
Median 5 min APGAR score [Median (Inter-Quartile Range); unit: Scores on a scale] — Appearance, Pulse, Grimace, Activity, and Respiration (APGAR), a 5-criteria assessment used to summarize the health of the newborn against infant mortality, scored at 5 minutes after birth. Each assessment (Appearance, Pulse, Grimace, Activity, and Respiration) is scored on a categorical scale of 0, 1 or 2 based on given criteria. All assessment scores are summarized to create the APGAR score (min = 0, max = 10). An APGAR score ≥7 generally indicates a newborn with normal health; An APGAR score ≤3 is generally considered critically low and cause for resuscitation efforts and critical care.
  Scores on a scale | 8 [7 to 8] | 7 [6 to 8] | 7 [7 to 8] | 7 [6 to 8] | 7 [7 to 8]

OUTCOME MEASURES:

1. Primary Outcome: Survival Without Evidence of Chronic Pulmonary Insufficiency of Prematurity (CPIP) at 12 Months Corrected Gestational Age (CGA)
Description: Number of events of survived participants without one or more of the CPIP components defined below:
  1. Medical/ER visits (CPIP-DV): At least one non-routine medical visit for respiratory causes.
  2. Respiratory re-hospitalizations (CPIP-RH): One or more re-hospitalizations for respiratory causes.
  3. Respiratory Symptoms (CPIP-SS): Evidence of respiratory symptoms (e.g. coughing and wheezing) or use of respiratory medications by parental diaries or pulmonary questionnaires.
  4. Respiratory Medications (CPIP-RM): Administration of respiratory medications (including oxygen).
  CPIP is defined as the presence of one or more parent-reported outcomes at 12 months CGA, validated by Respiratory diaries (presence of wheezing, coughing, and/or respiratory medication use ≥2 days per week for 3 consecutive weeks), and Pulmonary questionnaires (decrease in respiratory illness requiring medications, unscheduled medical visits and/or ER or hospital admissions).
Time Frame: 12 Months Corrected Gestational Age (*no imputation for missing data)
Population: Subjects were recruited from Tufts Medical Center, Brigham and Women's Hospital, Baystate Medical Center, Ginekologiczno-Położniczy Szpital Kliniczny Uniwersytetu Medycznego (UM), Instytut Centrum Zdrowia Matki Polski and Samodzielny Publiczny Zakład Opieki Zdrowotnej Szpital Uniwersytecki w Krakowie (USA, Poland).
Measure: Number; unit: Number of events
Units Other Than Participants: Number of events
Arm/Group | Placebo (Associated w/ Low Dose Cohort) | Low Dose (rhCC10) | Placebo (Associated w/ High Dose Cohort) | High Dose (rhCC10)
Number analyzed (Participants) | 22 | 22 | 21 | 23
Number analyzed (Number of events) | 41 | 25 | 33 | 29
Number of events
  Survived with no CPIP-DV (Medical/ER visits) | 8 | 2 | 6 | 6
  Survived with no CPIP-RH | 20 | 12 | 11 | 10
  Survived with no CPIP-SS (Respiratory Symptoms) | 2 | 3 | 6 | 5
  Survived with no CPIP-RM (Respiratory Medications | 10 | 7 | 6 | 5
  Survived with no CPIP events (-DV, -RH, -SS, -RM) | 1 | 1 | 3 | 3

2. Secondary Outcome: Long Term Efficacy - Survival Without Evidence of Chronic Pulmonary Insufficiency of Prematurity (CPIP) at 6 Months Corrected Gestational Age (CGA)
Description: Number of events of survived participants, graded as not having 1, 2, 3, or 4 of the CPIP components defined below:
  Medical/ER visits (CPIP-DV): ≥1 non-routine medical visit(s) for respiratory causes.
  Respiratory re-hospitalizations (CPIP-RH): ≥1 re-hospitalization(s) for respiratory causes Respiratory Symptoms (CPIP-SS): Parent-reported evidence of respiratory symptoms (e.g. coughing and wheezing) or use of respiratory medications Respiratory Medications (CPIP-RM): Administration of respiratory medications (including oxygen)
  A participant graded without 4 CPIP components is considered in better health than a participant graded without 1 CPIP component. CPIP components were parent-validated via respiratory diaries (wheezing, coughing, and/or respiratory medication use ≥2 days/wk for 3 consecutive wks), and pulmonary questionnaires (decrease in respiratory illness requiring medications, unscheduled medical visits and/or ER or hospital admissions).
Time Frame: 6 months Corrected Gestational Age
Population: Subjects were recruited from Tufts Medical Center, Brigham and Women's Hospital, Baystate Medical Center, Ginekologiczno-Położniczy Szpital Kliniczny UM, Instytut Centrum Zdrowia Matki Polski and Samodzielny Publiczny Zakład Opieki Zdrowotnej Szpital Uniwersytecki w Krakowie (USA, Poland).
Measure: Number; unit: Number of Events
Arm/Group | Placebo (Associated w/ Low Dose Cohort) | Low Dose (rhCC10) | Placebo (Associated w/ High Dose Cohort) | High Dose (rhCC10)
Number analyzed (Participants) | 22 | 22 | 21 | 23
Number of Events
  Survived without 1 CPIP component | 4 | 3 | 7 | 4
  Survived without 2 CPIP components | 10 | 6 | 8 | 7
  Survived without 3 CPIP components | 15 | 11 | 10 | 10
  Survived without 4 CPIP components | 21 | 16 | 17 | 14

3. Secondary Outcome: Safety and Efficacy - Number of Participants With Adverse Events
Description: The safety of the study drug was assessed by accounting the number of participants with Adverse Events (AEs) in the treatment and placebo groups.
Time Frame: Adverse events are monitored through 36 wks post-menstrual age (PMA)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (Associated w/ Low Dose Cohort) | Low Dose (rhCC10) | Placebo (Associated w/ High Dose Cohort) | High Dose (rhCC10)
Number analyzed (Participants) | 22 | 22 | 21 | 23
Participants | 22 | 22 | 21 | 23

4. Secondary Outcome: Short Term Efficacy - Number of Neonates With Oxygen Requirement at 36 Weeks Post Menstrual Age
Description: Short term efficacy evaluations involve number of neonates with oxygen requirement at 36 weeks post menstrual age.
Time Frame: 36 weeks post-menstrual age
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (Associated w/ Low Dose Cohort) | Low Dose rhCC10 | Placebo (Associated w/ High Dose Cohort) | High Dose rhCC10
Number analyzed (Participants) | 22 | 44 | 21 | 44
Participants | 8 | 10 | 8 | 4

ADVERSE EVENTS:
Time Frame: A given participant was monitored for Adverse Events (AE) and Serious Adverse Events (SAE) for an average of 34 months. Note: Some infants experienced the same AE on multiple occasions.
Description: AEs and SAEs were reported according to std. definitions, except AEs specific to this population and possibly relevant to the drug were automatically categorized as SAEs, regardless of severity, so each event would generate a report and be reviewed by study staff and the Data Safety and Monitoring Board (DSMB). AEs selected for automatic SAE reporting included; sepsis, pneumonia, air leaks (pneumothorax, pulmonary interstitial edema, pneumomediastinum), and pulmonary hemorrhage.
Arm/Group | Placebo (Associated w/ Low Dose Cohort) | Low Dose (rhCC10) | Placebo (Associated w/ High Dose Cohort) | High Dose (rhCC10)
All-Cause Mortality (participants affected / at risk) | 0/22 | 2/22 | 2/21 | 5/23
Serious Adverse Events (participants affected / at risk) | 16/22 | 17/22 | 17/21 | 19/23
Other Adverse Events (participants affected / at risk) | 22/22 | 22/22 | 21/21 | 23/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (Associated w/ Low Dose Cohort) (N=22) | Low Dose (rhCC10) (N=22) | Placebo (Associated w/ High Dose Cohort) (N=21) | High Dose (rhCC10) (N=23)
ROP Stage 3 (Eye disorders) | 5 (5) | 1 (1) | 3 (3) | 4 (4) — Retinopathy of prematurity
IVH grade 3-4 (Nervous system disorders) | 0 (0) | 1 (1) | 4 (4) | 4 (4) — Intraventricular Hemmorhage
PVL (Nervous system disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) — Periventricular leukomalacia
PDA (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 2 (2) | 3 (4) — Patent ductus arteriosus
Sepsis (Infections and infestations) | 1 (1) | 3 (3) | 3 (4) | 5 (6)
NEC Stage II-III (Gastrointestinal disorders) | 3 (3) | 1 (1) | 2 (2) | 2 (2) — Necrotizing enterocolitis
Intestinal Perforation (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (3) | 0 (0) | 4 (4)
Respiratory Acidosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Pulmonary Hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (2) | 2 (2)
Pulmonary Hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pulmonary Interstitial Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Apnea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 5 (5) | 1 (2) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1) | 0 (0) | 0 (0)
Respiratory Infections (Infections and infestations) | 5 (12) | 3 (4) | 9 (19) | 9 (17)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (Associated w/ Low Dose Cohort) (N=22) | Low Dose (rhCC10) (N=22) | Placebo (Associated w/ High Dose Cohort) (N=21) | High Dose (rhCC10) (N=23)
Apnea (Respiratory, thoracic and mediastinal disorders) | 22 (29) | 17 (22) | 10 (13) | 11 (12)
Anemia (Blood and lymphatic system disorders) | 10 (11) | 8 (9) | 16 (39) | 18 (50)
Pneumonia (Infections and infestations) | 3 (3) | 1 (1) | 8 (14) | 4 (11)
ROP Stages I-IV (Eye disorders) | 7 (11) | 2 (3) | 6 (7) | 8 (12) — Retnoipathy of Prematurity
IVH Grades I-IV (Nervous system disorders) | 3 (3) | 7 (7) | 9 (9) | 11 (11) — Intraventricular Hemmorhage
PVL Grades I-IV (Nervous system disorders) | 0 (0) | 0 (0) | 4 (4) | 0 (0) — Periventricular Leukomalacia
NEC Grades I-IV (Gastrointestinal disorders) | 3 (3) | 1 (1) | 4 (4) | 2 (2) — Necrotizing enterocolitis
Intestinal Perforation (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
PDA +ASD (Congenital, familial and genetic disorders) | 7 (7) | 9 (10) | 13 (14) | 14 (18) — Patent Ductus Arteriosus and Atrial Septal Defect
Sepsis (Infections and infestations) | 1 (1) | 3 (3) | 3 (4) | 5 (6)
UTI (Infections and infestations) | 2 (2) | 2 (2) | 3 (5) | 2 (3) — Urinary Tract Infection
Hyponatremia (Metabolism and nutrition disorders) | 4 (4) | 4 (4) | 2 (2) | 4 (5)
Metabolic Acidosis (Metabolism and nutrition disorders) | 8 (8) | 4 (4) | 6 (11) | 9 (12)
Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 1 (1) | 5 (5)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1) | 0 (0) | 1 (1)
Pulmonary Hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (2) | 2 (2)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
PIE (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 0 (0) | 1 (1) — Pulmonary Interstitial Emphysema
Bronchitis/ bronchiolitis/ tracheitis/laryngitis (Infections and infestations) | 7 (7) | 4 (6) | 2 (3) | 6 (6)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 1 (1) | 3 (3)
Respiratory Acidosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 4 (5) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 4 (4) | 3 (4) | 10 (10) | 8 (8)
Hypertension (Vascular disorders) | 2 (2) | 1 (1) | 1 (1) | 2 (2)
Hypotension (Vascular disorders) | 2 (3) | 2 (2) | 5 (6) | 9 (10)
Hernia (inguinal) (Gastrointestinal disorders) | 4 (4) | 3 (3) | 4 (6) | 3 (3)
Hyperbilirubinemia (Hepatobiliary disorders) | 15 (16) | 11 (11) | 11 (16) | 15 (20)
GERD (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1) | 5 (5)
Thrombocytopenia (Blood and lymphatic system disorders) | 4 (4) | 6 (6) | 5 (5) | 5 (6)
Thrombocytosis (Blood and lymphatic system disorders) | 0 (0) | 3 (3) | 0 (0) | 1 (2)
Desaturation after study medication administration (Investigations) | 4 (4) | 1 (1) | 1 (1) | 0 (0)
Coagulation disorders or circulatory insufficiency (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 4 (4) | 4 (4)
Hypoglycemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-10-01): https://cdn.clinicaltrials.gov/large-docs/45/NCT01941745/Prot_SAP_000.pdf